CLINICAL TRIAL: NCT01332227
Title: An Open-Label, Randomized Study Evaluating a Switch From a Regimen of Two Nucleoside Reverse Transcriptase Inhibitors Regimen Plus Any Third Agent to Either a Regimen of Atazanavir/Ritonavir Once Daily and Raltegravir Twice Daily or to a Regimen of Atazanavir/Ritonavir Once Daily and Tenofovir/Emtricitabine Once Daily in Virologically Suppressed HIV-1 Infected Subjects With Safety and/or Tolerability Issues on Their Present Treatment Regimen.
Brief Title: Atazanavir/Ritonavir, Once Daily + Raltegravir, Twice Daily, Switch Study in HIV-1-Infected Patients
Acronym: SPARTAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-402; 2009-017032-41 (EudraCT Number)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: HIV, Combination Therapy
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir; Raltegravir Potassium; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atazanavir/Ritonavir + Raltegravir (Experimental): Atazanavir + Ritonavir (heat-stable) + Raltegravir
  Interventions: Drug: Atazanavir; Drug: Ritonavir (heat-stable); Drug: Raltegravir
- Atazanavir/Ritonavir + Tenofovir/Emtricitabine (Other): Reference
  Atazanavir + Ritonavir (heat-stable) + Tenofovir/Emtricitabine
  Interventions: Drug: Atazanavir; Drug: Ritonavir (heat-stable); Drug: Tenofovir/Emtricitabine

INTERVENTIONS:
Drug: Atazanavir — Capsules, Oral, 300mg, Once daily, 48 weeks
  Other Names: Reyataz
Drug: Ritonavir (heat-stable) — Tablets, Oral, 100 mg, Once daily, 48 weeks
  Other Names: Norvir
Drug: Raltegravir — Tablets, Oral, 400 mg, Twice daily, 48 weeks
  Other Names: Isentress
  Arms: Atazanavir/Ritonavir + Raltegravir
Drug: Tenofovir/Emtricitabine — Tablets, Oral, 300/200 mg, Once daily, 48 weeks
  Other Names: Truvada
  Arms: Atazanavir/Ritonavir + Tenofovir/Emtricitabine

SUMMARY:
The purpose of this study is to determine whether HIV-1-infected patients, who are virologically suppressed on a regimen of 2 nucleoside reverse transcriptase inhibitors plus any third agent but are experiencing safety and/or tolerability issues, will maintain virologic suppression after switching to a regimen of heat-stable ritonavir boosted atazanavir, 300/100 mg, once daily plus raltegravir, 400 mg, twice daily.

DETAILED DESCRIPTION:
Allocation: Randomized nonstratified

Intervention model: Parallel versus comparator

ELIGIBILITY:
Key Inclusion Criteria

* Current treatment regimen of 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus any third agent for at least 3 months immediately prior to screening
* Virologic suppression (HIV-1 RNA <50 c/mL) for at least 3 months immediately prior to screening
* Virologic suppression (HIV-1 RNA <40 c/mL) using the Abbott m2000rt® polymerase chain reaction assay during screening period
* Treatment-related safety and/or tolerability issues to a regimen consisting of 2 NRTIs plus any third agent

Key Exclusion Criteria

* History of switch in highly active antiretroviral therapy due to virologic failure
* History of genotypic resistance to any component of the study regimen (atazanavir, raltegravir, tenofovir/emtricitabine)
* History of exposure to atazanavir/ritonavir or raltegravir prior to entering the study
* Experiencing safety and/or tolerability issues to tenofovir/emtricitabine or raltegravir
* Switch of any component of HIV antiretroviral medication regimen in the last 3 months immediately prior to or during the screening period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Mayers Squibb, Study Director — Bristol-Mayers Squibb
Locations (31):
- United States (8):
  - Health For Life Clinic Pllc, Little Rock, Arkansas
  - Eisenhower Medical Center, Palm Springs, California
  - Metropolis Medical Pc, San Francisco, California
  - Consultive Medicine, Daytona Beach, Florida
  - Orange County Health Dept., Orlando, Florida
  - Triple O Medical Services, P.A., West Palm Beach, Florida
  - The Research Institute, Springfield, Massachusetts
  - Aids Care, Rochester, New York
- France (5):
  - Local Institution, Paris, Cedex 12
  - Local Institution, Lyon
  - Local Institution, Orléans
  - Local Institution, Paris
  - Local Institution, Strasbourg
- Germany (5):
  - Local Institution, Bochum
  - Local Institution, Frankfurt
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
  - Local Institution, Munich
- Italy (3):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Roma
- Poland (2):
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Spain (3):
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Madrid
- United Kingdom (5):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Brighton
  - Local Institution, London
  - Local Institution, Sheffield

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 132 patients enrolled, 109 were randomized to receive treatment, and 23 patients were not randomized for the following reasons: 10 did not meet study criteria; 5 withdrew consent; 3 were lost to follow-up, and 5 withdrew for other reasons.
Groups:
- Atazanavir/Ritonavir + Raltegravir: Patients received atazanavir, 300-mg capsules, and ritonavir, 100-mg tablets, orally once daily and raltegravir, 400-mg tablets, twice daily for 48 weeks.
- Atazanavir/Ritonavir + Tenofovir/Emtricitabine: Patients received atazanavir, 300-mg capsules, plus ritonavir, 100-mg tablets, and tenofovir/emtricitabine, 300/200-mg tablets, orally once daily for 48 weeks.
Period: Overall Study
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Started | 72 (Participants who received treatment) | 37 (Participants who received treatment)
Completed | 56 | 32
Not Completed | 16 | 5
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lack of Efficacy | 3 | 1
Not completed — Poor compliance/noncompliance | 1 | 1
Not completed — Patient moved from area | 1 | 0
Not completed — Patient began prohibited medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine | Total
Number analyzed (Participants) | 72 | 37 | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] — Mean age
  Years | 43.1 (9.26) | 44.0 (10.38) | 43.4 (9.62)
Age, Continuous [Median (Full Range); unit: Years] — Median age
  Years | 44.0 [25 to 67] | 44.0 [25 to 69] | 44.0 [25 to 69]
Age, Customized [Number; unit: Participants]
  < 65 years | 69 | 36 | 105
  65-85 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 58 | 31 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 29 | 13 | 42
  Unknown or Not Reported | 38 | 23 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 54 | 24 | 78
  Black or African American | 8 | 6 | 14
  Hispanic | 2 | 0 | 2
  Unknown | 8 | 7 | 15
Mean CD4 count [Mean (Standard Deviation); unit: Cells/mm^3] | 587.7 (252.09) | 630.9 (270.02) | 601.5 (257.48)
Median CD4 count [Median (Full Range); unit: Cells/mm^3] | 588.5 [10 to 1511] | 639.5 [159 to 1395] | 593.0 [10 to 1511]
Cardiovascular disease risk factors [Number; unit: Participants] — Hypertension=systolic blood pressure/diastolic blood pressure >140/90 mm Hg or patient was taking antihypertensive medication; family history of coronary heart disease=father, mother, or sibling (male <55 years of age, and mother <65 years of age).
  Participants
    Hypertension | 5 | 6 | 11
    Diabetes mellitus | 3 | 1 | 4
    Current smoker | 27 | 11 | 38
    Previous smoker | 7 | 8 | 15
    Family history of premature coronary heart disease | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA Level <40 c/mL at Week 24
Description: HIV-1 RNA level was measured with the Abbott m2000rt® polymerase chain reaction assay. Response rates were assessed using an intent-to-treat algorithm, with numerator representing patients meeting the response criteria, and denominator representing all randomized patients. Randomized patients not meeting the criteria for treatment failure (eg, discontinuation of study therapy or virologic rebound at or before Week 24) were considered responders. Virologic rebound was defined as 2 consecutive on-treatment HIV-1 RNA levels ≥40 c/mL or the last on-treatment HIV-1 RNA level ≥40 c/mL followed by discontinuation. Patients who experienced treatment failure or had missing Week 24 HIV-1 RNA levels were considered failures. RNA=ribonucleic acid; HIV=human immunodeficiency virus.
Time Frame: From Day 1 to Week 24
Population: All patients who received study drug and who had an HIV-1 RNA measurement at the analysis week.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 72 | 37
Percentage of participants | 80.6 [69.5 to 88.9] | 94.6 [81.8 to 99.3]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA Level <40 c/mL at Week 48
Description: Percentages of patients with HIV-1 RNA levels <40 c/mL were summarized at each scheduled visit. Longitudinal plots were created to display proportion versus visit week through Weeks 24 and 48 with error bars representing 95% confidence intervals.
Time Frame: From Day 1 to Week 48
Population: All patients who received study drug and who had an HIV-1 RNA measurement at the analysis week.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 72 | 37
Percentage of participants | 69.4 [57.5 to 79.8] | 86.5 [71.2 to 95.5]

3. Secondary Outcome: Number of Participants With Virologic Rebound at Weeks 24 and 48
Description: Viral genotypic and phenotypic resistance profiles were assessed for virologic rebound (HIV-1 RNA level ≥40 c/mL). Only patients with HIV-1 RNA levels ≥500 c/mL met the criteria for resistance testing. Genotypic substitutions at baseline were summarized for virologic rebound. The genotypic resistance profile presented patients with genotypable isolates, those with protease inhibitor substitutions from genotypable isolates, those with integrase substitutions from genotypable isolates, and those with selected reverse transcriptase substitutions from genotypable isolates using the most current version of the International AIDS Society-USA list and Stanford HIV Drug Resistance Database. Newly emergent genotypic substitutions were summarized analogously for virologic rebound without baseline phenotypic resistance to atazanavir, ritonavir, or raltegravir, using all on-treatment isolates.
Time Frame: Day 1 to Weeks 28 and 48
Population: All patients who received study drug and who had an HIV-1 RNA measurement at the analysis week.
Measure: Number; unit: Participants
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 72 | 37
Participants
  Week 24: Virologic rebound | 7 | 1
  Week 48: Virologic rebound | 9 | 1

4. Secondary Outcome: Number of Participants With Genotypable/Phenotypable Isolates, Emergent Genotypic Substitutions in Patients With Genotypable Isolates, and Phenotypic Resistance in Patients With Phenotypable Isolates at Week 24
Description: Viral genotypic and phenotypic resistance profiles were assessed for virologic rebound (HIV-1 RNA level ≥40 c/mL). Only patients with HIV-1 RNA levels ≥500 c/mL met the criteria for resistance testing. Genotypic substitutions at baseline were summarized for virologic rebound. The genotypic resistance profile presented patients with genotypable isolates, those with protease inhibitor substitutions from genotypable isolates, those with integrase substitutions from genotypable isolates, and those with selected reverse transcriptase substitutions from genotypable isolates using the most current version of the International AIDS Society-USA list and Stanford HIV Drug Resistance Database. Newly emergent genotypic substitutions were summarized analogously for virologic rebound without baseline phenotypic resistance to atazanavir, ritonavir, or raltegravir, using all on-treatment isolates. pts=patients
Time Frame: Day 1 to Week 24
Population: Patients who received study drug, who had an HIV-1 RNA measurement at the analysis week and who experienced virologic rebound.
Measure: Number; unit: Participants
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 7 | 1
Participants
  Genotypable (GI)/phenotypable isolates (PI) | 4 | 0
  Emergent genotypic substitutions in GI pts (n=4,0) | 4 | 0
  Phenotypic resistance in PI pts (n=4,0) | 1 | 0

5. Secondary Outcome: Number of Participants With Genotypable/Phenotypable Isolates, Emergent Genotypic Substitutions in Patients With Genotypable Isolates, and Phenotypic Resistance in Patients With Phenotypable Isolates at Week 48
Description: as for outcome 4
Time Frame: Day 1 to Week 48
Population: Participants with virologic rebound
Measure: Number; unit: Participants
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 9 | 1
Participants
  Genotypable (GI)/phenotypable isolates (PI) | 5 | 0
  Emergent genotypic substitutions in GI pts (n=5,0) | 5 | 0
  Phenotypic resistance in PI pts (n=5,0) | 1 | 0

6. Secondary Outcome: Number of Patients With Death as Outcome, Serious Adverse Events (SAEs), Treatment-related SAEs, Treatment-emergent Adverse Events (AEs) Leading to Discontinuation, and Treatment-emergent AEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug.
Time Frame: Day 1 to Week 48
Population: All participants who received study drug
Measure: Number; unit: Particpants
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 72 | 37
Particpants
  Deaths | 0 | 0
  SAEs | 4 | 1
  Related SAEs | 1 | 0
  Treatment-emergent AEs leading to discontinuation | 3 | 1
  Treatment-emergent AEs | 51 | 28

7. Secondary Outcome: Mean Changes in Fasting Lipid Levels From Baseline to Week 48
Description: LD=low-density lipoprotein; HDL=high-density lipoprotein.
Time Frame: From Baseline to Week 48
Population: All participants who received study drug
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Number analyzed (Participants) | 72 | 37
mg/dL
  Fasting total cholesterol | 11.7 (5.239) | -10.2 (4.769)
  Fasting LDL cholesterol | 7.7 (3.986) | -5.4 (4.691)
  Fasting HDL cholesterol | 2.7 (2.055) | -0.3 (1.915)
  Fasting non-HDL cholesterol | 9.0 (4.983) | -9.8 (4.430)
  Fasting triglycerides | 14.7 (16.667) | -17.6 (16.994)

ADVERSE EVENTS:
Arm/Group | Atazanavir/Ritonavir + Raltegravir | Atazanavir/Ritonavir + Tenofovir/Emtricitabine
Serious Adverse Events (participants affected / at risk) | 4/72 | 1/37
Other Adverse Events (participants affected / at risk) | 27/72 | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir/Ritonavir + Raltegravir (N=72) | Atazanavir/Ritonavir + Tenofovir/Emtricitabine (N=37)
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir/Ritonavir + Raltegravir (N=72) | Atazanavir/Ritonavir + Tenofovir/Emtricitabine (N=37)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 4 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Ocular icterus (Eye disorders) | 6 | 3
Gonorrhoea (Infections and infestations) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 4
Headache (Nervous system disorders) | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Bronchitis (Infections and infestations) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.